CLINICAL TRIAL: NCT00068276
Title: Orthomolecular Vitamin D3 in Low-Risk Myelodysplastic Syndrome: An Open-Label Clinical Trial
Brief Title: Cholecalciferol in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU-29203; CDR0000318802 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-BG03-117
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: previously treated myelodysplastic syndromes; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: cholecalciferol

SUMMARY:
RATIONALE: Cholecalciferol (vitamin D) may improve quality of life by increasing blood counts, decreasing fatigue, and improving other symptoms of myelodysplastic syndrome.

PURPOSE: This phase II trial is studying how well cholecalciferol works in treating patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of cholecalciferol, in terms of hematological improvement, in patients with low- or intermediate-risk myelodysplastic syndromes.
* Determine the effect of this drug on disease symptoms, fatigue, and the overall health-related quality of life of these patients.

OUTLINE: This is an open-label, pilot study.

Patients receive oral cholecalciferol once daily. Treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed myelodysplastic syndromes (MDS)

  * Must have undergone bone marrow aspirate and biopsy with karyotype within the past 3 months
* International Prognostic Scoring System score of 0 or 1

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Any

Life expectancy

* More than 1 year

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* No history of hypercalcemia

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior stem cell transplantation allowed
* No concurrent hematopoietic growth factors

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 6 weeks since prior cholecalciferol supplements or analogs
* More than 4 weeks since any prior therapy for MDS (except supportive care)
* No other concurrent therapy for MDS

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2005-06 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Molnar, MD, Study Chair — Wake Forest University Health Sciences; Bayard L. Powell, MD — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina, United States